CLINICAL TRIAL: NCT07361757
Title: Qualia Perimenopause Efficacy and Tolerability Study: An Open-label 3-Arm Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qualia Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: QLS-022
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Peri-menopausal Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Qualia Perimenopause Formula A (Experimental)
  Interventions: Dietary Supplement: Qualia Perimenopause Formula A
- Qualia Perimenopause Formula B (Experimental)
  Interventions: Dietary Supplement: Qualia Perimenopause Formula B
- Qualia Perimenopause Formula C (Experimental)
  Interventions: Dietary Supplement: Qualia Perimenopause Formula C

INTERVENTIONS:
Dietary Supplement: Qualia Perimenopause Formula A — Qualia Perimenopause is a multi-botanical natural health product/dietary supplement formulated to support women during the perimenopausal transition. The formulation is intended to address common domains of symptom burden-including vasomotor, psychological, cognitive, and sleep-related complaints-through complementary mechanisms of action. Participants receive one capsule once daily for 28 consecutive days. Three different formulations are being tested in this trial (Formula A, Formula B, and Formula C).
  Arms: Qualia Perimenopause Formula A
Dietary Supplement: Qualia Perimenopause Formula B — Qualia Perimenopause is a multi-botanical natural health product/dietary supplement formulated to support women during the perimenopausal transition. The formulation is intended to address common domains of symptom burden-including vasomotor, psychological, cognitive, and sleep-related complaints-through complementary mechanisms of action. Participants receive one capsule once daily for 28 consecutive days. Three different formulations are being tested in this trial (Formula A, Formula B, and Formula C).
  Arms: Qualia Perimenopause Formula B
Dietary Supplement: Qualia Perimenopause Formula C — Qualia Perimenopause is a multi-botanical natural health product/dietary supplement formulated to support women during the perimenopausal transition. The formulation is intended to address common domains of symptom burden-including vasomotor, psychological, cognitive, and sleep-related complaints-through complementary mechanisms of action. Participants receive one capsule once daily for 28 consecutive days. Three different formulations are being tested in this trial (Formula A, Formula B, and Formula C).
  Arms: Qualia Perimenopause Formula C

SUMMARY:
This is an open-label, 3-arm clinical trial evaluating the short-term efficacy and tolerability of Qualia Perimenopause-a multi-ingredient dietary supplement formulated to support perimenopausal symptoms-in healthy women aged 40-55 who are symptomatic but not yet menopausal (menses within the past 12 months). Approximately 120 participants will be allocated across three parallel arms and will take 1 capsule once daily for 28 consecutive days. The primary outcome is between-group change from baseline to day 28 in menopause symptom burden measured by the total Menopause Rating Scale (MRS). Secondary outcomes include within- and between-group changes at days 14 and 28 in cognitive function (PROMIS Cognitive Function v2.0 - Short Form 8a), sleep disturbance (PROMIS), MRS subdomains (psychological, somato-vegetative, urogenital), overall MRS change, safety/tolerability (custom survey), and participant-reported product experience. All assessments are completed electronically at home at baseline, mid-intervention (day 14), and end-of-study (day 28), with a brief follow-up questionnaire; there are no in-person visits.

DETAILED DESCRIPTION:
Perimenopause is a transitional phase preceding menopause characterized by fluctuating ovarian hormone levels and variable cycle length, often accompanied by a constellation of symptoms spanning vasomotor disturbances, sleep disruption, cognitive and attentional changes, mood lability, somatic complaints, and urogenital discomfort. These symptoms can meaningfully impair quality of life, productivity, interpersonal functioning, and health-related well-being. Although menopausal hormone therapy is an established option for selected individuals, many women either do not elect or are not candidates for hormone-based interventions and seek nonhormonal approaches that address multiple symptom domains concurrently. In this context, multi-ingredient botanical formulations are of growing interest as supportive strategies designed to target the diverse and interrelated pathways implicated in perimenopausal symptomatology.

Qualia Perimenopause is a multi-botanical natural health product/dietary supplement formulated to support women during the perimenopausal transition. The formulation is intended to address common domains of symptom burden-including vasomotor, psychological, cognitive, and sleep-related complaints-through complementary mechanisms of action.

Study Design: This is an open-label, three-arm, parallel-group trial with stratified randomization by baseline Menopause Rating Scale (MRS) total score. Participants will be stratified and randomly assigned to one of three study arms in a 1:1:1 ratio. Study duration is 28 days of supplementation.

Participants will take one capsule once daily of their assigned formula for 28 consecutive days. All data are self-reported; assessments are completed electronically at home at baseline, mid-intervention (day 14), and end-of-study (day 28), with a brief follow-up questionnaire. Approximately 120 healthy female participants ages 40-55 with menopause symptoms but not yet in menopause (period within last 12 months) and MRS total score ≥ 5 will be enrolled.

ELIGIBILITY:
Inclusion criteria:

1. Provide voluntary, written, informed consent to participate in the study
2. Agree to provide a valid cell phone number and are willing to receive communications through text
3. Can read and write English
4. Willing to not begin taking any new supplements during the study and continue taking any supplements they are currently using regularly
5. Willing to complete questionnaires, records, and diaries associated with the study
6. Healthy female participants ages 40-55 with menopause symptoms but not yet in menopause (period within last 12 months)
7. MRS total score ≥ 5 (preference given to higher score)

Exclusion criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant or start breastfeeding during the trial
2. Known food intolerances/allergy to any ingredients in the product
3. Having any of the following conditions: Psychiatric conditions, neurologic disorders, endocrine disorders, cancer
4. Having had a significant cardiovascular event in the past 6 months
5. Taking MAO inhibitors, SSRIs, or any other psychiatric or neurological medicines
6. On immunosuppressive therapy
7. Having had surgery within the past 6 weeks or upcoming planned surgery in the next few months
8. Adults lacking capacity to consent
9. Post-menopause (≥12 consecutive months without a period)
10. Taking medications: hormone replacement therapy; oral contraceptives; selective estrogen receptor modulators/aromatase inhibitors (e.g., Tamoxifen); sedatives/anxiolytics; blood thinners; insulin

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Menopause Rating Scale (MRS) - Total Score | Day 28
  Between-group change from baseline to Day 28 in menopause symptoms measured by the total Menopause Rating Scale (MRS) score. The MRS is an 11-item self-rating scale that measures the severity of menopausal symptoms with a total score range of 0-44.

SECONDARY OUTCOMES:
PROMIS Cognitive Function v2.0 - Short Form 8a | Day 14, Day 28
  Within- and between-group changes from baseline to Days 14 and 28 in cognitive function measured by PROMIS Cognitive Function v2.0 - Short Form 8a, an 8-item assessment of perceived cognitive abilities including mental acuity, concentration, and memory.
Safety and Tolerability Survey | Day 14, Day 28
  Within- and between-group changes from baseline to Days 14 and 28 in side effect profile using a custom Safety and Tolerability survey assessing symptoms including nausea, headache, mood changes, dizziness, bloating, itching, and sexual dysfunction.
PROMIS Sleep Disturbance - Short Form | Day 14, Day 28
  Within- and between-group changes from baseline to Days 14 and 28 in sleep measured by PROMIS Sleep Disturbance - Short Form, an 8-item assessment of sleep quality, restfulness, and disturbance severity.
MRS Psychological Subdomain | Day 14, Day 28
  Within- and between-group changes from baseline to Days 14 and 28 in the Psychological subdomain of the Menopause Rating Scale (items 4-7: depressive mood, irritability, anxiety, exhaustion).
MRS Somato-Vegetative Subdomain | Day 14, Day 28
  Within- and between-group changes from baseline to Days 14 and 28 in the Somato-vegetative subdomain of the Menopause Rating Scale (items 1-3, 11: hot flashes, heart discomfort, sleep problems, joint/muscle discomfort).
MRS Urogenital Subdomain | Day 14, Day 28
  Within- and between-group changes from baseline to Days 14 and 28 in the Urogenital subdomain of the Menopause Rating Scale (items 8-10: sexual problems, bladder problems, vaginal dryness).
Follow-up Questionnaire | Day 33 (5-7 days after final dose)
  Participant thoughts and feelings about the product assessed via a Follow-up Questionnaire administered 5-7 days after the final dose. Evaluates overall experience, product rating, purchase interest, and detailed product experience description.

IPD SHARING:
Plan to Share IPD: No